CLINICAL TRIAL: NCT04037813
Title: Comparative Study of Hysteroscopic Versus Laparoscopic Tubal Occlusion in Cases of Communicating Hydrosalpinx and Planning for IVF
Brief Title: Hysteroscopic Versus Laparoscopic Tubal Occlusion in Cases of Hydrosalpinx and Planning for IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Abdel Salam, Assistant lecturer in obstetrics and gynecology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140689
Record Dates: First submitted 2019-07-21; First posted 2019-07-30 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Tubal Obstruction
Keywords: Hysteroscopy; Laparoscopy; Hydrosalpinx
MeSH Terms: conditions — Fallopian Tube Diseases | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic tubal occlusion (Active Comparator): 54 patients will undergo laparoscopic tubal occlusion.
  Interventions: Procedure: Laparoscopic and hysteroscopic tubal occlusion for hydrosalpinx
- Hysteroscopic tubal occlusion (Active Comparator): 54 patients will undergo hysteroscopic tubal occlusion.
  Interventions: Procedure: Laparoscopic and hysteroscopic tubal occlusion for hydrosalpinx

INTERVENTIONS:
Procedure: Laparoscopic and hysteroscopic tubal occlusion for hydrosalpinx — For hysteroscopic tubal occlusion group it will be done under general anesthesia using standard, rigid 4-mm hysteroscopy with a 30° forward-oblique lens and a 5.5-mm diagnostic sheath (Karl Storz , Germany). Uterine distension allowed a panoramic view of the uterine cavity and identification of the tubal ostia.The roller ball (Ball Electrode, unipolar, 5 Fr) will be used for the coagulation of the interstitial part of the tube and the uterine cornu area.
  For laparoscopic tubal occlusion group it will be done under general anesthesia using bipolar coagulation and a proximal tubal cut.

SUMMARY:
compare the efficacy of hysteroscopic tubal occlusion versus laparoscopic tubal occlusion for the patients of communicating hydrosalpinx scheduled for IVF. half of the patients will undergo hysteroscopic tubal occlusion while the other half will undergo laparoscopic tubal occlusion.

DETAILED DESCRIPTION:
The study will include 108 patients complaining of infertility associated with unilateral or bilateral tubal communicating hydrosalpinx. All the patients will be subjected to informed consent, history taking, full physical examination, ultrasound examination via transvaginal approach using ultrasound machine ( Voluson Pro-V and GE Voluson E 10) and HSG within the last 6 months showing unilateral or bilateral communicating hydrosalpinx.

The patients (108) will be equally randomized into two groups :

Group (A): 54 patients (Hysteroscopic tubal occlusion group). Group (B): 54 patients (Laparoscopic tubal occlusion group). Randomization will be done using 108 opaque sealed envelopes that will be numbered serially from 1-108 and each envelope corresponding letter which denotes the allocated group will be put according to randomization table then all envelopes will be closed and put in one box, when the first patient arrives, after giving informed consent, the first envelope will be opened and the patient will be allocated according to the letter inside.

For hysteroscopic tubal occlusion group it will be done under general anesthesia using standard, rigid 4-mm hysteroscopy with a 30° forward-oblique lens and a 5.5-mm diagnostic sheath (Karl Storz , Germany). Uterine distension allowed a panoramic view of the uterine cavity and identification of the tubal ostia.The roller ball (Ball Electrode, unipolar, 5 Fr) will be used for the coagulation of the interstitial part of the tube and the uterine cornu area.

For laparoscopic tubal occlusion group it will be done under general anesthesia using bipolar coagulation and a proximal tubal cut. The contraindications for laparoscopy were mainly extensive abdominal or pelvic adhesions of various etiologies (e.g. previous surgery, pelvic inflammatory disease, and pelvic endometriosis) and morbid obesity.

The operative details of hysteroscopic tubal occlusion and laparoscopic tubal occlusion including operative time and complications will be documented In both groups, the patients will be followed up for the next 24 hours as regard post-operative pain (using VAS ) and post-operative recovery (patient mobilization, intestinal motility and patient discharge).

The success rate of tubal occlusion will be assessed one month later using post-menstrual HSG and for hysteroscopic group office hysteroscopy will be done for assessment of uterine cavity after electrocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility.
* The presence of communicating hydrosalpinx diagnosed by HSG,TV U/S showing distended tubes and intrauterine fluid or patient complaining of prolonged brownish vaginal discharge.
* Candidate for IVF procedure.

Exclusion Criteria:

* Uterine anomalies.
* Serious medical condition and unfit for surgery.
* Contraindication for laparoscopic tubal occlusion.
* Contraindication for pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with successful hysteroscopic tubal occlusion | one month post-operative.
  Successful tubal occlusion will be measured by the presence of negative spill and proximal tubal block on HSG.

SECONDARY OUTCOMES:
The percentage of patients with successful laparoscopic tubal occlusion | one month post-operative.
  Successful tubal occlusion will be measured by the presence of negative spill and proximal tubal block on HSG.
The post-operative pain in both groups (using VAS ). | 24 hours post-operative.
  The patients will be followed up for the next 24 hours as regard post-operative pain (using VAS) .
The operative time and complications in both groups. | Intra-operative duration.
  the operative time and operative complications will be documented according to the hospital records .
Compare the success rate of tubal occlusion in both groups. | one month post-operative.
  The number of HSG that showed post-operative tubal occlusion in hysteroscopic group compared to laparoscopic group.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Abdelsalam, Msc, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No